CLINICAL TRIAL: NCT02986659
Title: Genomic Outcomes of Metformin
Acronym: GOMET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB00034977
Record Dates: First submitted 2016-10-27; First posted 2016-12-08 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease; Mild Cognitive Impairment; Obesity, Abdominal; Hypertension
MeSH Terms: conditions — Coronary Artery Disease; Cognitive Dysfunction; Obesity, Abdominal; Hypertension | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin then Placebo (Active Comparator): Metformin dosing at 425, 850 and 1700 mg with GLUCOPHAGE® (metformin hydrochloride) Tablets. Treatment with metformin will be initiated at a dose of 425 mg (half pill) taken orally once a day at night for 7 days. After the week, the participant will be called to assess tolerance and will be asked to increase dose to one pill at night at a dose of 850 mg for one week. At the end of the second week, participants will be called again and if they tolerated the second dose, they will be asked to take two 850 mg pills, one in the morning and one at night, for a total dose of 1700 mg which is within the range of the usual effective dose of 1500 to 2000 mg/day for the remainder of the 3 months. Will then cross over to 3 months on placebo.
  Interventions: Drug: Metformin; Drug: Placebo
- Placebo then Metormin (Placebo Comparator): Dietary Supplement: Placebo with Methylcellulose capsules. Treatment with placebo will be initiated at a dose of a half pill taken orally once a day at night for 7 days. After the week, the participant will be called to assess tolerance and will be asked to increase dose to one pill at night for one week. At the end of the second week, participants will be called again and if they tolerated the second dose, they will be asked to take two pills, one in the morning and one at night for the remainder of the 3 months. After 3 months on placebo, participants will then cross over to 3 months of metformin as described in the other arm.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin
Drug: Placebo

SUMMARY:
Medical scientists have found that people with diabetes who take the drug Metformin have less age-related disease than those taking other treatments and researchers believe it may prevent numerous diseases and conditions that effect older people. In addition, metformin extends lifespan in some animal models of human disease. The purpose of this study is to see if taking Metformin causes changes in blood cells consistent with improved health and longevity in people who do not have diabetes. In this study Metformin will be compared to placebo. A placebo is a substance, like a sugar pill, that is not thought to have any effect on a participants disease or condition. In this study participants will either receive the active study medication, Metformin or placebo which is not active. Placebos are used in research studies to see if the drug being studied really does have an effect.

DETAILED DESCRIPTION:
The number of older adults is projected to increase dramatically by 2050. Aging-related diseases and conditions still seriously compromise the quality of life among most older adults. Several pharmaceutical agents, such as metformin, have been tested to extend lifespan and delay aging-related diseases and dysfunctions in mice. Metformin, a biguanide antidiabetic drug, reduces the risk for developing type-2 diabetes in persons at risk by over one-third with few adverse effects (e.g., gastrointestinal irritation). Metformin prevents type-2 diabetes primarily through decreasing hepatic glucose synthesis, as well as enhancing insulin sensitivity and increasing peripheral glucose uptake. The molecular mechanisms remain unclear, although a number of potential mechanism such as activation of AMP-activated protein kinase (AMPK) and inhibition of mitochondrial glycerophosphate dehydrogenase have been proposed. The fact that metformin treatment in persons with type-2 diabetes has been associated with reduced risk of other aging-related diseases and conditions, including cardiovascular disease, cancer and cognitive decline supports the possibility of the beneficial effects of metformin on healthy aging. It is imperative to capitalize on these leads to extend health span among older adults.

To translate animal findings to human intervention trials, appropriate aging biomarkers are needed. Methylomic and transcriptomic profiles in relevant cells may reflect molecular features that mediate effects of both genetic and environmental factors on aging-related functional decline and disease. The roles of monocytes have been implicated in development of many aging-related diseases such as cardiovascular disease, cancer and neurodegenerative disease. In a cross-sectional association study of 1,200 monocyte samples, we identified 1,794 age-associated methylation sites and 2,704 age-associated transcripts, which were over-represented in two networks (autophagy and oxidative phosphorylation) and suggestive of decline in those functions with age. Both autophagy and oxidative phosphorylation are considered as key contributors to the aging process, and their dysfunctions have been linked to aging-related diseases. Changes in these aging-related omic biomarkers may be early indicators of cellular damage or disruption that eventually leads to age-related dysfunctions. Assessment of these aging biomarkers in response to therapeutic intervention may also provide molecular insight for personalizing treatment. The investigators propose a pilot study to examine changes in aging-related omic profiles after 3 months of metformin treatment in 35 monocyte samples from older adults using a randomized, double-blind, placebo-controlled crossover study design.

Our overarching goal of the pilot study is to evaluate the utility of using the aging-related omic biomarkers as an indicator of pharmacologic responses in the anti-aging therapeutic intervention trials through the following specific aims. Although this pilot study does not have sufficient power to definitively test all the aims, it will provide essential preliminary data for developing a full scale research program.

* Aim 1A: To test the effects of the metformin treatment on transcriptomic profiles and related functional changes in human monocytes,
* Aim 1B: To explore the effects of the metformin treatment on methylomic profiles in human monocytes,
* Aim 2: To investigate the longitudinal relationship between transcriptional and functional changes in human monocytes during the metformin treatment and
* Aim 3: To test the effects of the metformin treatment on frailty and other aging-related physical and cognitive measures and investigate the longitudinal relationship between these changes and transcriptional changes.

A randomized, double-blind, placebo-controlled crossover trial in 30 participants using metformin and matching placebo will be used. In the absence of a treatment by sequence interaction effect, this design can increase study power for evaluating treatment effects by allowing each participant to be his/her own control. The period effect may be minimum because the primary outcomes, methylation and transcriptional measures, are relatively stable overtime.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 79

Must meet criteria from one or more of the following groups:

Group 1 (Can have 1 or 2 of these, but not all 3)

* History of coronary artery disease (MI/heart attack, stroke, heart failure, or peripheral artery disease)
* Cancer, with no active treatment in the last year
* MCI (MoCA >18<26 -inclusive of 1 point if <12 years of education Group 2
* Decline physical function (walking speed < 1 m/s) Group 3 (Either or both)
* Abdominal obesity (>88cm women, >102cm men) AND hypertension (treated or resting blood pressure >140/90
* Abdominal obesity (>88cm women, >102cm men) AND hyperlipidemia (treated or fasting total cholesterol >240 English literacy Willing to provide informed consent

Exclusion Criteria:

* eGFR <45
* Type 2 diabetes (HbA1c>6.5) or type 1 diabetes
* Any tobacco or nicotine product use in the past year
* Low vitamin B12 Levels (< 300 pg/mL)
* Self-reported severe difficulty or inability to walk 400m or climb 10 steps (from Q 2 and 19 on PAT-D)
* Self-reported difficulty or inability to perform basic ADL functions (from Q 10, 13, 14, 16 on PAT-D)
* Excessive alcohol use (>14 drinks/week)
* Cancer requiring treatment in past year (except skin)
* Dementia - diagnosed and/or MoCA score <18
* Parkinson's or other neurological disease
* Chronic liver disease or cirrhosis
* End stage renal disease or on dialysis
* Rheumatic conditions (Rheumatoid arthritis, lupus, and any other autoimmune disease the -PI deems them to be ineligible for)
* Thyroid problems the PI deems them to be ineligible for
* Gout
* Involved in another interventional study
* Hemoglobin <8 or diagnosed with anemia
* Recent unintentional weight change (+/- 10 lbs. in the last 12 months)
* BMI <18.5
* Likely to not follow the protocol
* PI deems unfit to participate
* Already taking Metformin or any other drug intended to treat diabetes

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jingzhong Ding, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin Then Placebo: Metformin dosing at 425, 850 and 1700 mg with GLUCOPHAGE® (metformin hydrochloride) Tablets. Treatment with metformin will be initiated at a dose of 425 mg (half pill) taken orally once a day at night for 7 days. After the week, the participant will be called to assess tolerance and will be asked to increase dose to one pill at night at a dose of 850 mg for one week. At the end of the second week, participants will be called again and if they tolerated the second dose, they will be asked to take two 850 mg pills, one in the morning and one at night, for a total dose of 1700 mg which is within the range of the usual effective dose of 1500 to 2000 mg/day for the remainder of the 3 months. Will then cross over to 3 months on placebo.
  Metformin
  Placebo
- Placebo Then Metormin: Dietary Supplement: Placebo with Methylcellulose capsules. Treatment with placebo will be initiated at a dose of a half pill taken orally once a day at night for 7 days. After the week, the participant will be called to assess tolerance and will be asked to increase dose to one pill at night for one week. At the end of the second week, participants will be called again and if they tolerated the second dose, they will be asked to take two pills, one in the morning and one at night for the remainder of the 3 months. After 3 months on placebo, participants will then cross over to 3 months of metformin as described in the other arm.
  Metformin
  Placebo
Period: First Intervention Period
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Started | 15 | 15
Completed | 11 | 13
Not Completed | 4 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention Period
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Started | 11 | 13
Completed | 11 | 7
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin Then Placebo | Placebo Then Metormin | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Total number of patients enrolled was 30, but 7 patients did not complete at least one of the two intervention periods. Numbers in baseline analysis includes only the subjects who completed.
  years
    number analyzed (Participants) | 11 | 12 | 23
    (all) | 71.07 (3.58) | 71.67 (4.13) | 71.4 (3.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total number of patients enrolled was 30, but 7 patients did not complete at least one of the two intervention periods. Numbers in baseline analysis includes only the subjects who completed.
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    Female | 6 | 7 | 13
    Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number of patients enrolled was 30, but 7 patients did not complete at least one of the two intervention periods. Numbers in baseline analysis includes only the subjects who completed.
  Participants
    number analyzed (Participants) | 11 | 12 | 23
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 11 | 12 | 23
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Eigengene Scores
Description: Part of blood sample analysis will give results for Individual methylation sites and transcripts, especially the eigengenes of autophage, oxidative phosphorylation and protein synthesis networks Methylomic and transcriptomic profiles in monocytes. All of the results for these measures will be aggregated into an eigengene score. The eigengene score is a summary measure of a group of correlated genes. This score may indicate status of a biological function. In this analysis, the observed range of values were from -0.48 to 0.66. A lower score means downregulation of the gene group, while a higher score upregulation. No theoretical minimum or maximum value exist for this assay.
Time Frame: baseline through 12 weeks
Population: Numbers differ from baseline due to subject withdraw or lost to follow up
Measure: Mean (Standard Deviation); unit: Eigen Score
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 11 | 12
Eigen Score | .035 (.24) | -0.032 (.35)

2. Primary Outcome: Change in Eigengene Scores
Description: as for outcome 1
Time Frame: baseline through 24 weeks
Population: Numbers differ from baseline due to subject withdraw or lost to follow up
Measure: Mean (Standard Deviation); unit: Eigen Score
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 10 | 6
Eigen Score | .011 (.28) | -0.018 (.36)

3. Secondary Outcome: Functional Measures--macroautophagy
Description: Macroautophagy is a process of wrapping cellular components inside autophagosomes and delivering them to lysosomes for degradation.
Time Frame: baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Measures--microautophagy
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Functional Measures--chaperone-mediated Autophagy
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mitochondria Function: Respiratory Control Ratio (RCR)
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mitochondria Function: State 3 (Maximal Oxygen Consumption Rate)
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mitochondria Function: State 4 (Oxygen Consumption Upon Inhibition of ATP Synthase)
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Population: Unable to collect and analyze these measures due to lack of funding--samples were not collected.
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Vital Signs
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Expanded Short Physical Performance Battery (eSPPB)
Description: Score ranges from 0 (low physical function) to 12 (high physical function).
Time Frame: From baseline through 12 weeks
Population: Changes in population due to withdraw/loss to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 11 | 12
score on a scale | .45 (.82) | .27 (1.35)

11. Other Pre Specified Outcome: Change in Expanded Short Physical Performance Battery (eSPPB)
Description: Score ranges from 0 (low physical function) to 12 (high physical function).
Time Frame: From 12 weeks through 24 weeks
Population: Changes in population due to withdraw/loss to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 10 | 6
score on a scale | -.010 (0.74) | 0.00 (0.63)

12. Other Pre Specified Outcome: Nottingham Power Rig
Description: The Nottingham power rig evaluates mean unilateral leg muscle power
Time Frame: Baseline through 12 weeks, 12 weeks through 24 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Grip Strength
Description: measurement of the amount of static force that the hand can squeeze
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: Change in score. Score ranges from 0 (low cognitive function) to 30 (high cognitive function).
Time Frame: Baseline through 12 weeks
Population: Changes in participant numbers are due to due to withdraw/loss to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 11 | 12
score on a scale | -0.091 (2.02) | 0.91 (1.22)

15. Other Pre Specified Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: Change in score. Score ranges from 0 (low cognitive function) to 30 (high cognitive function).
Time Frame: 12 weeks through 24 weeks
Population: Changes in participant numbers are due to due to withdraw/loss to follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metformin Then Placebo | Placebo Then Metormin
Number analyzed (Participants) | 10 | 6
score on a scale | 1.90 (1.60) | 0.50 (1.38)

16. Other Pre Specified Outcome: Blood Lipids--total Cholesterol
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Blood Lipids--HDL-Cholesterol
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Blood Lipids--Triglycerides
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Blood Lipids--calculated LDL Levels
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Mobility Assessment Tool - Short Form (MAT-sf).
Description: MAT-sf is a tool for assessing self-perception of mobility. The possible range of score is from 30 to 80 with lower score indicating lower perception of mobility.
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Pepper Assessment Tool for Disability (PAT-D)
Description: The PAT-D is a self-administered questionnaire which consists of 23 items that include a range of activities that assess mobility, activities of daily living (ADL) and instrumental activities of daily living (IADL). Responses are made on a five-point Likert scale ranging from 1 ("usually did with no difficulty") to 5 ("unable to do") or a box can be checked that reads "usually did not do for other reasons".
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Medication Adherence
Description: Amount of medication expected to be taken vs. amount participant actually takes.
Time Frame: Baseline through 12 weeks and 12 weeks through 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through week 24
Groups:
- Metformin: Metformin dosing at 425, 850 and 1700 mg with GLUCOPHAGE® (metformin hydrochloride) Tablets. Treatment with metformin will be initiated at a dose of 425 mg (half pill) taken orally once a day at night for 7 days. After the week, the participant will be called to assess tolerance and will be asked to increase dose to one pill at night at a dose of 850 mg for one week. At the end of the second week, participants will be called again and if they tolerated the second dose, they will be asked to take two 850 mg pills, one in the morning and one at night, for a total dose of 1700 mg which is within the range of the usual effective dose of 1500 to 2000 mg/day for the remainder of the 3 months.
- Placebo: Placebo will be given for 3 months.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=30) | Placebo (N=30)
Gastrointestinal--Nausea/Diarrhea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Itching (General disorders) | 1 (1) | 0 (0)
Palpitation (Cardiac disorders) | 1 (1) | 0 (0)
Ataxia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT02986659/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02986659/ICF_001.pdf